CLINICAL TRIAL: NCT00883454
Title: Estimation of Functional Liver Reserve in Patients With Hepatocellular Carcinoma in Cirrhosis: the Value of Preoperative Cholinesterases
Brief Title: Estimation of Functional Liver Reserve Using Cholinesterases
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Other Study IDs: CHE-HCC
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Last update posted 2009-04-17 (Estimated); Status verified 2009-04

CONDITIONS: Hepatocellular Carcinoma; Cirrhosis; Liver Neoplasm; Liver Disease
Keywords: hepatocellular carcinoma; liver tumor; cirrhosis; liver resection; tumor staging; liver disease staging
MeSH Terms: conditions — Carcinoma, Hepatocellular; Fibrosis; Liver Neoplasms; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Estimation of functional liver reserve in patients with hepatocellular carcinoma (HCC) in cirrhosis is of paramount importance to properly select candidates for surgical resection. Together with the value of bilirubin, the presence/absence of ascites and esophageal varices, and the rate of residual liver volume, which are our current parameters to measure functional liver reserve, the investigators sought to investigate the value of preoperative cholinesterases (CHE) in predict postoperative adverse outcome after hepatic resection for HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Total bilirubin < 2 mg/dl
2. No ascites
3. No esophageal varices, or esophageal varices eradicated by endoscopy
4. Liver volume:

   * residual liver volume > or = 40% if total bilirubin < 1 mg/dl
   * residual liver volume > or = 50% if total bilirubin between 1 and 1.5 mg/dl
   * only limited resection if total bilirubin > 1.5 mg/dl
5. Portal vein embolization was selected in any case in whom RLV did not fit the previous requirements.

Exclusion Criteria:

1. Total bilirubin > 2 mg/dl
2. Refractory ascites
3. Esophageal varices

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The records of approximately 245 consecutive patients who were referred at our Unit because of HCC were reviewed. Among those, 191 (78%) were submitted to surgery, and 181 (74%) were resected. The patients excluded from surgery were addressed to symptomatic treatments because of advanced disease or impaired liver functional reserve, or to percutaneous ablation therapy according to our policy. Among resected patients, there were 145 (80%) men and 36 (20%) women, with median age of 67 years (range 36-87 years).
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)

PRIMARY OUTCOMES:
The primary outcome was to investigate the value of preoperative cholinesterases in predict postoperative adverse outcome after hepatic resection for hepatocellular carcinoma in cirrhosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Liver Surgery Unit, Third Department of Surgery, University of MIlan, IRCCS Istituto Clinico Humanitas, Rozzano, Milan, Milan, Italy